CLINICAL TRIAL: NCT06712953
Title: The Effect of Repeated Standardized Patient Use on Students' Anxiety and Learning Levels in Teaching Extremity Examination Skills
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Suleyman Demirel University (Other)
Responsible Party: Principal Investigator, Tuğçe Çamlıca, Lecturer, Dr, Suleyman Demirel University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 72867572-050.01.04-616349
Record Dates: First submitted 2024-11-26; First posted 2024-12-03 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: Nursing Students
Keywords: Anxiety; self-confidence; active learning; passive learning; psychomotor skills; standardized patient; peer; extremity
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- the peer assessment group (Experimental): Students in the peer assessment group were paired (by randomization, on their request) to have a teammate of the same sex before the extremity examination experience. In the following process, the students were asked to perform extremity examinations in line with the specified objectives.
  Interventions: Other: the peer assessment group
- the standardized patient group (Experimental): Students in the standardized patient group were asked to perform extremity examinations per the specified objectives in standardized patient.
  Interventions: Other: the peer assessment group

INTERVENTIONS:
Other: the peer assessment group — Students in the peer assessment group were paired (by randomization, on their request) to have a teammate of the same sex before the extremity examination experience. In the following process, the students were asked to perform extremity examinations in line with the specified objectives. Students in the standardized patient group were asked to perform extremity examinations per the specified objectives in standardized patient.

SUMMARY:
Aims: This study aimed to examine the effects of peer assessment and repeated standardized patient use on students' self-confidence and anxiety and their psychomotor skill performance in teaching extremity examination skills.

Design: This randomized controlled experimental study was carried out following the CONSORT checklist.

Methods: The study sample consisted of second-grade nursing students enrolled in the " Health Diagnosis" course in the fall semester of the 2023-2024 academic year (n:67). The students in the peer assessment group performed the upper and lower extremity examinations once whereas those in the standardized patient group performed these examinations three times. Research data were analyzed in IBM SPSS 25.0 (Statistical Package for Social Sciences) software. The Shapiro-Wilk test was used to check whether the data were normally distributed. Parametric and nonparametric tests and descriptive statistical methods were used for data analysis. The significance levels were taken as p<0.001 and p<0.05. The scales used were analyzed with the Cronbach alpha reliability coefficient; the scenarios and forms created by the researchers were evaluated with the Lawshe Technique.

ELIGIBILITY:
Inclusion Criteria:

* Second-grade nursing students
* Enrolled in the " Health Diagnosis" course at the Faculty of Health Sciences, Department of Nursing of a university in the fall semester of the 2023-2024 academic year

Exclusion Criteria:

- Students who actively continue their nursing profession as well as their education life

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2023-11-09 (Actual); Primary Completion 2023-12-21 (Actual); Study Completion 2023-12-21 (Actual)

PRIMARY OUTCOMES:
Extremity examinations | First week
  The students in the standardized patient group performed extremity examinations on the same standardized patient three times, whereas the students in the peer assessment group performed this examination on their peers once

OTHER OUTCOMES:
First measurement (Self-conficent and Anxiety) | First week
  The students in the standardized patient group performed extremity examinations on the same standardized patient three times, whereas the students in the peer assessment group performed this examination on their peers once.
Second measurement (Self-conficent and Anxiety) | Third week
  The students in the standardized patient group performed extremity examinations on the same standardized patient three times, whereas the students in the peer assessment group performed this examination on their peers once
Third measurement (Self-conficent and Anxiety) | fifth week
  The students in the standardized patient group performed extremity examinations on the same standardized patient three times, whereas the students in the peer assessment group performed this examination on their peers once

CONTACTS AND LOCATIONS:
Locations (1):
- Suleyman Demirel University, Isparta, Center, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Aydin AG, Ince S. The effect of Jigsaw technique on nursing students' psychomotor skill levels and academic achievement: A quasi-experimental study. Nurse Educ Pract. 2023 Nov;73:103821. doi: 10.1016/j.nepr.2023.103821. Epub 2023 Oct 30. PMID 37952472